CLINICAL TRIAL: NCT00598858
Title: Phase II Study to Determine the Effects of Neoadjuvant Docetaxel on Newly Diagnosed Intermediate and High Grade Cancer of the Prostate in Patients Who Are Scheduled for Radical Prostatectomy With Genomic Correlates of Pathological Response
Brief Title: Neoadjuvant Docetaxel on Newly Diagnosed Intermediate and High Grade Cancer of the Prostate
Acronym: 2007-5904
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted due to zero accrual and lack of funding
Sponsor: John P. Fruehauf (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, John P. Fruehauf, Dr. John P. Fruehauf, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 07-14; 2007-5904 (Other: University of California, Irvine); NCI-2012-02085 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate; Stage I Prostate Cancer; Stage II Prostate Cancer
Keywords: prostate cancer; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (docetaxel and prednisone) (Experimental): Patients receive docetaxel IV over 60 minutes on days 1 and 2 and prednisone PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: 114977-28-5; 40466; 628503; RP 56976; RP56976; Taxotere; TXT
Drug: Prednisone — Given PO
  Other Names: Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta(1)-Cortisone; Delta-Dome; Deltacortene; deltacortisone; deltadehydrocortisone; Deltison; Deltra; Econosone; Liquid Pred; Lisacort; Meprosona-F; metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRD; PRED; Predeltin; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; Sk-Prednisone; Sterapred

SUMMARY:
This pilot phase II trial studies docetaxel and prednisone in treating patients with newly diagnosed stage I-II prostate cancer undergoing prostatectomy. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as prednisone, may stimulate the immune system in different ways and stop cancer cells from growing. Giving docetaxel and prednisone together may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of a 3-month prostate-specific antigen (PSA) decline of at least 30% by chemotherapy regimen of docetaxel and prednisone in patients with stage I/II prostate cancer, who are scheduled for prostatectomy.

II. To compare tumor, pathological and PSA responses to neoadjuvant docetaxel between patients with intermediate and high grades of prostate cancer.

III. To obtain prostate specimens for genomic correlates with responses of the chemotherapy regimen of docetaxel and prednisone.

OUTLINE:

Patients receive docetaxel intravenously (IV) over 60 minutes on days 1 and 2 and prednisone orally (PO) twice daily (BID) on days 1-21. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients undergo prostatectomy within 3 weeks after completion of chemotherapy.

After completion of study treatment, patients are followed up within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histological diagnosis of adenocarcinoma of the prostate which is measurable or evaluable Stage I or II.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patient must have a pre-study PSA within 28 days prior to start of therapy.
* Patients who have received prior radiotherapy are not eligible.
* Patient must have an adequate renal function
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Age > 18
* Patients must be able to take oral medications

Exclusion Criteria:

* Patients with measurable metastatic diseases by a CT scan of the abdomen and pelvis within 28 days and by a bone scan within 42 days prior to start of therapy.
* Patient must not have received chemotherapy, biologic therapy or any other investigational drug for any reason within 28 days prior to start of therapy and must have recovered from toxicities of prior therapy to grade 1 or less with the exception of alopecia.
* Patients must not be treated with non-steroidal anti-androgens (flutamide, bicalutamide, nilutamide or ketoconazole).
* Patients must not take vitamins, herbs, or micronutrient supplement within 28 days prior to start of therapy.
* Patients may not have ongoing problems with bowel obstruction or short bowel syndrome characterized by grade 2 or greater diarrhea or malabsorptive disorders.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Patients should not have psychological, familial, sociological, or geographical conditions that do not permit medical follow-up or compliance with the study protocol.
* Patients should not have any medical life-threatening complications of their malignancies
* Patients should not have a known severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, active uncontrolled infection, or HIV).
* Patients should not have current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Patients with history of myocardial infarction, cerebrovascular accident, transient ischemic attack, or unstable angina within 6 months
* Patients with clinically significant peripheral vascular disease
* Patients with evidence of bleeding diathesis or coagulopathy
* Patients with central nervous system or brain metastases
* Patients who had major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Patients with minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Patients with history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
* Patients with serious, non-healing wound, ulcer, or bone
* Patients who are diagnosed of any other malignancy except non-melanomatous skin cancer in the past 5 years
* Patients receiving anticoagulation therapy (e.g. Coumadin) prior to registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PSA response rate (partial response (PR) + complete response (CR)) | 9 weeks
  Expressed with two-sided exact binomial confidence intervals. Significance of changes between pre- and after-treatment PSA or testosterone will be determined by the Wilcoxon signed-rank test. The difference of response rates between different pre-treatment pathological stages or Gleason scores will also be examined by Fisher's exact test. Associations between PSA response and tumor response, and PSA response and gene expression will also be examined by Fisher's exact test.

SECONDARY OUTCOMES:
Rates of tumor response | Up to 7 days after completion of study treatment
  Expressed with two-sided exact binomial confidence intervals.
The rate of negative surgical margin | Up to 7 days after completion of study treatment
The proportion of patients with pathological down-staging defined as evidence of decreased pathological stage or Gleason score when compared with pretreatment pathological stage | Up to 7 days after completion of study treatment
Adverse events defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment | Up to 28 days after completion of study treatment
  Severity will be categorized by toxicity grade according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: John P. Fruehauf, MD, PhD, Principal Investigator — University of California, Irvine